CLINICAL TRIAL: NCT02046005
Title: Communication of Biomarker, Genetic, and Lifestyle Risk Factor Profiles for Rheumatoid Arthritis to First Degree Relatives
Brief Title: Personalized Risk Estimator for Rheumatoid Arthritis Family Study
Acronym: PRE-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Elizabeth Karlson, M.D., Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P60 AR047782-6121; P60AR047782 (NIH)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: First Degree Relatives of Rheumatoid Arthritis Patients
Keywords: Family History; RA; Rheumatoid Arthritis; Genetics; Rheumatoid Factor; Shared Epitope; Anti-CCP
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- General Rheumatoid Arthritis Education (Active Comparator): Arm 1 participants will receive general information about RA.
  Interventions: Behavioral: General Rheumatoid Arthritis Education
- PRE-RA (Experimental): Arm 2 participants will receive personalized RA risk education by the PRE-RA risk tool.
  Interventions: Behavioral: PRE-RA
- PRE-RA Plus (Experimental): Arm 3 participants will receive personalized RA risk education by the PRE-RA risk tool and health educator.
  Interventions: Behavioral: PRE-RA Plus

INTERVENTIONS:
Behavioral: PRE-RA — Personalized Risk Estimator for Rheumatoid Arthritis (PRE-RA) is an online tool that provides education about RA, collects data about demographics and behaviors, and presents personalized RA risk information.
  Other Names: Personalized Risk Estimator for RA
  Arms: PRE-RA
Behavioral: PRE-RA Plus — Personalized Risk Estimator for Rheumatoid Arthritis (PRE-RA) is an online tool that provides education about RA, collects data about demographics and behaviors, and presents personalized RA risk information. In addition, participants in this arm receive education from a health educator.
  Other Names: Personalized Risk Estimator for RA with Health Educator
  Arms: PRE-RA Plus
Behavioral: General Rheumatoid Arthritis Education — Participants will receive general information about signs and symptoms of rheumatoid arthritis.
  Arms: General Rheumatoid Arthritis Education

SUMMARY:
The purpose of this study is to understand how personalized risk factors for rheumatoid arthritis (RA) may impact willingness to change behaviors associated with RA. The investigators have developed a personalized risk estimator for RA based on demographics, family history, biomarkers and behaviors related to RA risk. Eligible participants have a first degree relative with RA but do not have RA themselves. Participants who meet eligibility and consent to the study will be randomized to receive either standard information about RA, the online personalized RA risk tool, or the online personalized RA risk tool with guidance from a health educator. Participants will be followed to measure willingness to change RA risk behaviors. The investigators hypothesize that participants who receive the online personalized RA risk tool and health education will be more willing to change RA risk behaviors compared to participants that receive standard RA information.

DETAILED DESCRIPTION:
A risk tool for rheumatoid arthritis (RA) was developed to provide personalized risk communication that includes biomarker, genetic and lifestyle RA risk factors. This risk calculator is referred to as the Personalized Risk Estimator for Rheumatoid Arthritis (PRE-RA) which will be used in the PRE-RA Family Study. A 3-arm randomized trial will be conducted among 222 RA first degree relatives that will be followed for one year. Participants will be surveyed before and after RA education concerning (i) knowledge and attitudes about RA risk, (ii) decisional balance related to behaviors, and (iii) stage of behavior change concerning lifestyle risks.

At the initial study visit, participants will be randomly assigned to one of three arms. Arm 1 participants will receive general education about RA (comparison group). These participants will be followed to assess for willingness to change behaviors associated with RA risk. Arm 2 participants will receive personalized risk by the personalized RA risk tool (PRE-RA). These participants will be followed to assess for willingness to change RA risk behaviors. Arm 3 participants will receive personalized risk by the online risk tool along with health education and counseling (PRE-RA Plus group). These participants will be followed to assess for willingness to change RA risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* First degree blood relative (parent, sibling, or child) with diagnosis of RA
* Age between 18 and 70 years old

Exclusion Criteria:

* Non-English speaking
* Sign/symptoms of rheumatoid arthritis (assessed by screening questionnaire and study staff)
* Rheumatoid arthritis
* Systemic lupus erythematosus
* Juvenile Idiopathic Arthritis
* Psoriatic Arthritis
* Ankylosing Spondylitis
* Mixed Connective Tissue Disease
* Reactive Arthritis
* Adult-Onset Still's Disease
* Sjogren's Syndrome
* Dermatomyositis
* Polymyositis
* Polymyalgia Rheumatica
* ANCA-associated Vasculitis
* Giant Cell Arteritis
* Polyarteritis Nodosa
* Behcet's Disease
* Relapsing Polychondritis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W Karlson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sparks JA, Iversen MD, Miller Kroouze R, Mahmoud TG, Triedman NA, Kalia SS, Atkinson ML, Lu B, Deane KD, Costenbader KH, Green RC, Karlson EW. Personalized Risk Estimator for Rheumatoid Arthritis (PRE-RA) Family Study: rationale and design for a randomized controlled trial evaluating rheumatoid arthritis risk education to first-degree relatives. Contemp Clin Trials. 2014 Sep;39(1):145-57. doi: 10.1016/j.cct.2014.08.007. Epub 2014 Aug 20. PMID 25151341
- [Result] Sparks JA, Iversen MD, Yu Z, Triedman NA, Prado MG, Miller Kroouze R, Kalia SS, Atkinson ML, Mody EA, Helfgott SM, Todd DJ, Dellaripa PF, Bermas BL, Costenbader KH, Deane KD, Lu B, Green RC, Karlson EW. Disclosure of Personalized Rheumatoid Arthritis Risk Using Genetics, Biomarkers, and Lifestyle Factors to Motivate Health Behavior Improvements: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Jun;70(6):823-833. doi: 10.1002/acr.23411. Epub 2018 Apr 16. PMID 29024454
- [Derived] Prado MG, Iversen MD, Yu Z, Miller Kroouze R, Triedman NA, Kalia SS, Lu B, Green RC, Karlson EW, Sparks JA. Effectiveness of a Web-Based Personalized Rheumatoid Arthritis Risk Tool With or Without a Health Educator for Knowledge of Rheumatoid Arthritis Risk Factors. Arthritis Care Res (Hoboken). 2018 Oct;70(10):1421-1430. doi: 10.1002/acr.23510. PMID 29316383

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General Rheumatoid Arthritis Education | PRE-RA | PRE-RA Plus
Started | 80 | 78 | 80
Completed | 72 | 71 | 70
Not Completed | 8 | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Rheumatoid Arthritis Education | PRE-RA | PRE-RA Plus | Total
Number analyzed (Participants) | 80 | 78 | 80 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (14.7) | 45.0 (14.9) | 48.3 (13.7) | 45.6 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 62 | 57 | 182
  Male | 17 | 16 | 23 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 65 | 73 | 207
  Non-White | 11 | 13 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Contemplation Ladder
Description: Measures willingness to change any of 4 RA-related behaviors compared to baseline using generalized estimating equations to compare the PRE-RA groups to the comparison arm.
Time Frame: Immediately, 6 weeks, and 6 months after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | General Rheumatoid Arthritis Education | PRE-RA | PRE-RA Plus
Number analyzed (Participants) | 80 | 78 | 80
Participants
  Immediately post-intervention | 40 | 46 | 43
  6 weeks post-intervention | 41 | 49 | 45
  6 months post-intervention | 40 | 53 | 48
Statistical Analysis 1: Comparison: General Rheumatoid Arthritis Education vs PRE-RA vs PRE-RA Plus; In the primary analysis, we combined the PRE-RA and PRE-RA Plus arms into a single "PRE-RA group" and compared it to the Comparison arm (aka "General Rheumatoid Arthritis Education"); Test type: Superiority; p = 0.043, generalized estimating equations — We compared the PRE-RA group (PRE-RA arm and PRE-RA Plus arm combined) to the Comparison arm for the primary composite outcome at the 3 primary post-intervention time points using generalized estimating equations (GEE); Risk Ratio (RR) = 1.23, 95% CI 2-sided [1.01 to 1.51] — PRE-RA group (combined PRE-RA arm and PRE-RA Plus arm) compared to Comparison arm (reference)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Behavioral intervention
Arm/Group | General Rheumatoid Arthritis Education | PRE-RA | PRE-RA Plus
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/78 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/78 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/78 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No